CLINICAL TRIAL: NCT07298941
Title: An Adaptive Intervention to Improve Pain Outcomes Following Cognitive Behavioral Therapy for Insomnia in Patients With Comorbid Chronic Low Back Pain and Insomnia
Brief Title: Resilience Enhancement Following Sleep Treatment
Acronym: REST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Patrick Finan, PhD, Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SBS-7457; R01AT013240 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain (CLBP); Insomnia
Keywords: chronic low back pain; insomnia; cognitive-behavioral therapy for insomnia; meditation; savoring; pain; internet intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Adaptive Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-Behavioral Therapy for Insomnia (Other): Open Label CBTi
  Interventions: Behavioral: Cognitive-behavioral therapy for insomnia (CBTi)
- Cognitive-Behavioral Therapy for Insomnia plus Savoring Meditation (Experimental): Open label CBTi followed by random allocation to Savoring Meditation
  Interventions: Behavioral: CBTi + Savoring Meditation
- Cognitive-Behavioral Therapy for Insomnia plus Pain Education (Active Comparator): Open label CBTi followed by random allocation to Pain Education
  Interventions: Behavioral: CBTi + Pain Education

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy for insomnia (CBTi) — Sleep Healthy Using the Internet (SHUTi) is a 9-week self-guided, automated, internet-based program that is tailored to the individual and designed to recapitulate the core features of face-to-face CBTi (sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, relapse prevention). It is fully accessible as a web-based application via computers, tablets, and smartphones.
  Arms: Cognitive-Behavioral Therapy for Insomnia
Behavioral: CBTi + Savoring Meditation — After first completing CBTi, participants will then complete a course of Savoring Meditation, a meditation training program focused on generating and maintaining positive emotions. Savoring Meditation training comprises four 30-minute training sessions (20-minute meditation training and 10 minutes for Q&A and session debrief), and will be delivered 1-on-1 by a trained interventionist over remote video-conference.
  Arms: Cognitive-Behavioral Therapy for Insomnia plus Savoring Meditation
Behavioral: CBTi + Pain Education — After first completing the full course of CBTi, participants will then complete a Pain Education intervention. Delivered 1-on-1 via telehealth, patients will be introduced to the biopsychosocial model of pain, through which they will learn about 1) biological bases for low back pain and chronic pain in general, 2) psychological and 3) social processes that influence pain perception, and 4) pain self-management strategies that are supported by scientific evidence. Pain Education training comprises four 30-minute training sessions.
  Arms: Cognitive-Behavioral Therapy for Insomnia plus Pain Education

SUMMARY:
The primary objective of this study is to evaluate the efficacy of an adaptive intervention targeting both insomnia and positive affect in improving pain outcomes for adults with chronic low back pain (cLBP) and comorbid insomnia. Specifically, the study tests whether augmenting a cognitive behavioral therapy for insomnia (CBTi) program with a meditation intervention (Savoring Meditation) or a Pain Education intervention will result in greater reductions in pain intensity.

Secondary objectives include evaluating improvements in insomnia severity, positive and negative affect, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

(1) age >=18 years; (2) report low back pain as ongoing problem >= 3 months and any pain on at least half of the days over the past 6 months (consistent with NIH Consensus Recommendations, other chronic pain problems can be present, but cLBP must be reported as primary); (3) average pain intensity >= 4 over past 7 days on a 0-10 numerical rating scale; (4) sleep-onset insomnia and/or sleep maintenance insomnia and/or late insomnia (>30 minutes of WASO or SOL or waking >30 minutes before desired time for at least 3 nights/week) with presence of insomnia symptoms for >= 6 months, and the sleep disturbance (or associated daytime fatigue) must cause significant distress or impairment in social, occupational, or other areas of functioning to be consistent with DSM 5 criteria (evaluated by phone interview).

Exclusion Criteria:

(1) currently receiving behavioral treatment for insomnia; (2) currently engaging in formal or informal meditation practice on a regular (e.g., weekly) basis; (3) unstable medication use for sleep, pain, or other indication (e.g., changed within the past 3 months); (4) irregular sleep schedules dictated by shift work (i.e., usual bedtimes outside 8:00 p.m.-2:00 a.m. or arising time outside 4:00 a.m.-10:00 a.m.); (4) mental health condition deemed to interfere with study procedures or put the participant at undue risk via semi-structured interview (e.g., screen positive for psychotic disorder) or other untreated sleep disorders (e.g., obstructive sleep apnea, restless legs syndrome) as evaluated by our semi-structured interview based on the Diagnostic Interview for Insomnia (DII); (5) do not have regular internet access; (6) cannot read and speak English (interventions only available in English); and (7) severe cognitive impairment (i.e., score =9 on the Telephone-Assessed Mental State); (8) currently pregnant; 9) unable or unwilling to comply with study protocols, or otherwise determined by the PI to be able to safely participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | Baseline to post-intervention (11 weeks)
  0-10 pain severity item from the PEG

SECONDARY OUTCOMES:
Pain Severity | Baseline to 6 months follow-up
  0-10 pain severity item from the PEG
Pain Severity | Baseline to 12 month follow-up
  0-10 pain severity item from the PEG
Pain Interference | Baseline to Post-Intervention (11 weeks), 6 month follow-up, 12 month follow-up
  Pain interference items from the PEG
Disability | Baseline to Post-Intervention (11 weeks), 6 month follow-up, 12 month follow-up
  Oswestry Disability Index
Insomnia Severity | Baseline to Post-Intervention (11 weeks), 6 month follow-up, 12 month follow-up
  Insomnia Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Finan, Ph.D., Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will consider data sharing requests on a case by case basis, as dictated by institutional data sharing agreements.